CLINICAL TRIAL: NCT02490514
Title: Mircera In Patients With CKD Stages III-IV Not On Dialysis: Observational, Non-interventional Cohort Study
Brief Title: A Study Of Mircera In Patients With Kidney Disease Who Are Not On Dialysis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25065
Record Dates: First submitted 2015-07-02; First posted 2015-07-03 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Renal Tubular Acidosis, Distal, With Hemolytic Anemia
MeSH Terms: conditions — Renal Tubular Acidosis, Distal, With Hemolytic Anemia

STUDY DESIGN:
Observational Model: Cohort

GROUPS / COHORTS (1):
- Mircera: Patients with stage III-IV CKD received open-label Mircera for 12 months at a dose to be determined by the investigator.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention was administered in this study.

SUMMARY:
This open-label, non-randomized, retrospective-prospective, non-interventional study will evaluate the efficacy and safety of Mircera in patients with stage III-IV chronic kidney disease (CKD) not on dialysis. Patients will receive open-label treatment with Mircera for 12 months at a dose to be determined by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage II-IV CKD not on dialysis, including renal transplant patients, who are receiving erythropoiesis-stimulating agent (ESA) treatment or are ESA-naive
* Patients who will not require dialysis within 12 months after the start of Mircera therapy
* Patients whose life expectancy is greater than 12 months after Mircera initiation
* Patients >/= 18 years and </= 75 years of age
* Patients who are female and of childbearing potential must be using effective contraception methods
* Patients with no contra-indications to ESA treatment (for example, hypersensitivity, non-controlled hypertension and others according to the local SmPC)
* Patients who have given written informed consent where local regulations allow or require it

Exclusion Criteria:

* Patients with stage I-II or stage V CKD
* Poorly controlled hypertension
* Active malignant disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 to 75 years old with stage III-IV chronic kidney disease not on dialysis
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2009-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Percent Of Participants Who Reached And Maintained Target Hemoglobin Values During Treatment | 12 months

SECONDARY OUTCOMES:
Hb Levels At Start And End Of Treatment | 12 months
Mircera Dose At Start And End Of Treatment | 12 months
Time To Achieve Response To Mircera | 12 months
Percent Of Participants Treated With Iron Supplements | 12 months
Percent of Participants Who Required Transfusion At Start And End Of Treatment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- Serbia (10):
  - Belgrade
  - Ćuprija
  - Kragujevac
  - Niš
  - Pirot
  - Požarevac
  - Sremska Mitrovica
  - Šabac
  - Užice
  - Zrenjanin